CLINICAL TRIAL: NCT00382291
Title: SSRI-Induced Activation Syndrome in Pediatric Obsessive Compulsive Disorder
Brief Title: Effectiveness of Sertraline and Cognitive Behavioral Therapy in Treating Pediatric Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: R01MH078594 (NIH); R01MH078594 (NIH); DSIR 84-CTM
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2012-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Antidepressive Agents, Second-Generation; Placebos; Cognitive Behavior Therapy; Child Psychiatry; Activation Syndrome; Psychometrics
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Regular Titration (Experimental): Regular titration of Sertraline plus cognitive behavioral therapy. The titration schedule used a flexible upward titration from 25 mg/day to 200 mg/day over 9 weeks unless higher doses were not tolerated, after which the dosage was adjusted as a function of tolerability. If tolerated, maximum dose could be achieved in 5 weeks.
  Interventions: Drug: Regular Titration
- Placebo (Placebo Comparator): Placebo plus cognitive behavioral therapy
  Interventions: Drug: Placebo
- Slow Titration (Experimental): Slow titration of Sertraline plus cognitive behavior therapy. The titration schedule utilized a slower titration schedule relative to the RegSert arm. Unless unable to tolerate higher doses, children remained on 25mg/day for the first two weeks, 50mg/day from weeks 3-4, 75mg/day for weeks 5-6, 100mg/day for week 7, 150mg/day for week 8, and 200mg/day for week 9 until the end of the study.
  Interventions: Drug: Slow Titration

INTERVENTIONS:
Drug: Regular Titration — Sertraline will be administered in standard dosing. Treatment with sertraline will last 18 weeks.
  Arms: Regular Titration
Drug: Placebo — The placebo will be administered in the same manner as sertraline. Treatment with placebo will last 18 weeks.
  Arms: Placebo
Drug: Slow Titration — Sertraline will be administered in slow titration. Treatment with sertraline will last 18 weeks.
  Arms: Slow Titration

SUMMARY:
This study measures the occurrence of certain side effects linked to antidepressant use and evaluates the effectiveness of the medication sertraline plus cognitive behavioral therapy to treat people with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is an anxiety disorder that is associated with recurring repetitive behaviors and persistent unwanted thoughts. People with OCD often carry out ritual-like behaviors such as counting, cleaning, or washing their hands in order to momentarily ease their anxiety. A current treatment for people with OCD is the class of antidepressants called selective serotonin reuptake inhibitors (SSRIs). A recent re-analysis of clinical trials on children with psychiatric conditions found that the risk of suicidal thoughts and behavior when on SSRI-antidepressants was considerably higher than when on placebo. The data also revealed that antidepressant-associated suicidal behavior was not limited to children with depression, but also affected children with OCD and other anxiety disorders. Although the process responsible for increased suicidality is unknown, it may be initiated by a set of symptoms collectively called SSRI induced activation syndrome, which is thought to be common, particularly in children and teens. However, there is a lack of knowledge on this syndrome, including its role in suicidal behavior and how it can be prevented. This study will evaluate a new behavioral test to measure certain side effects linked to antidepressant use. This study will also evaluate the effectiveness of the SSRI sertraline plus cognitive behavioral therapy (CBT) to treat people with OCD.

Potential participants will undergo an initial screening visit that will include an interview on psychological symptoms associated with OCD and possible family history of OCD. Eligible participants will then undergo a physical exam, blood draw, DNA sampling, and pregnancy test if applicable. Participants will be randomly assigned to receive either sertraline or placebo daily for 18 weeks. At weekly study visits, participants will receive their study drug, complete questionnaires about symptoms of OCD, and undergo vital sign measurements. At specified visits, participants will also perform a task (Stop Signal Task) on a computerized assessment device to measure attention and impulse control and may have blood drawn. For the first 4 weeks participants will wear a wristwatch-like device (actigraph) to monitor sleep patterns. During the first three visits, participants will receive supportive psychotherapy. At Visit 4, participants will begin receiving 60-minute CBT sessions, which will continue until the final visit. The final visit will include a second physical exam, questionnaires, and blood testing.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of OCD with at least a 6-month duration, as determined by structured clinical interview (schedule for affective disorders and schizophrenia for school-age children)
* As long as OCD is the principal diagnosis, co-morbid depression, attention deficit hyperactivity disorder, tic disorder, or another anxiety disorder is allowable
* Diagnosis of trichotillomania or body dysmorphic disorder provided OCD symptoms are the predominant presenting features
* Meets clinical criteria for Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal Infections (PANDAS) (e.g., abrupt onset and dramatic fluctuations in symptoms)

Exclusion Criteria:

* Prior adequate trial of sertraline
* Allergy to sertraline
* History of rheumatic fever or serious autoimmune disorder
* Diagnosis of bipolar disorder, autism, schizophrenia, mental retardation, or chronic degenerative neurological disease
* Current anorexia nervosa with symptoms of body image distortion (symptoms of anorexia secondary to obsessions [e.g., contamination] are permitted)
* Unable to safely swallow study medication after pill swallowing education
* Unwillingness of children's parents to commit to accompanying their child for multiple study visits and to be responsible for medication compliance
* Suicidal intent (suicidal ideation will not be an automatic exclusion; however, risk will be gauged carefully and the participant must contract for safety)
* Suicide attempt in the 12 months prior to study entry
* Pregnancy
* Taking monoamine oxidase inhibitors (MAOIs) within 4 weeks of study entry or fluoxetine within 5 weeks of study entry
* Taking other psychotropic medications other than sedative or hypnotics for insomnia
* Substance abuse or dependence within 6 months prior to study entry

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya K. Murphy, MD, Principal Investigator — University of South Florida; Regina Bussing, M.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida

REFERENCES:
- [Result] Bussing R, Murphy TK, Storch EA, McNamara JP, Reid AM, Garvan CW, Goodman WK. Psychometric properties of the Treatment-Emergent Activation and Suicidality Assessment Profile (TEASAP) in youth with OCD. Psychiatry Res. 2013 Feb 28;205(3):253-61. doi: 10.1016/j.psychres.2012.09.019. Epub 2012 Sep 29. PMID 23031804
- [Derived] Reid AM, McNamara JP, Murphy TK, Guzick AG, Storch EA, Goodman WK, Geffken GR, Bussing R. Side-effects of SSRIs disrupt multimodal treatment for pediatric OCD in a randomized-controlled trial. J Psychiatr Res. 2015 Dec;71:140-7. doi: 10.1016/j.jpsychires.2015.10.006. Epub 2015 Oct 14. PMID 26495770
- [Derived] Bussing R, Reid AM, McNamara JP, Meyer JM, Guzick AG, Mason DM, Storch EA, Murphy TK. A pilot study of actigraphy as an objective measure of SSRI activation symptoms: results from a randomized placebo controlled psychopharmacological treatment study. Psychiatry Res. 2015 Feb 28;225(3):440-5. doi: 10.1016/j.psychres.2014.11.070. Epub 2014 Dec 10. PMID 25535011
- [Derived] Storch EA, Bussing R, Small BJ, Geffken GR, McNamara JP, Rahman O, Lewin AB, Garvan CS, Goodman WK, Murphy TK. Randomized, placebo-controlled trial of cognitive-behavioral therapy alone or combined with sertraline in the treatment of pediatric obsessive-compulsive disorder. Behav Res Ther. 2013 Dec;51(12):823-9. doi: 10.1016/j.brat.2013.09.007. Epub 2013 Oct 10. PMID 24184429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at two child and adolescent psychiatric clinics within university medical centers: Gainesville, Florida (FL) (UF) and Tampa, FL (USF). Recruitment started in early 2009 and ended in late 2010.
Pre-assignment Details: Fifteen participants were excluded after screening: 7/15 did not meet inclusion/exclusion criteria and 8/15 withdrew consent.
Groups:
- Placebo Plus CBT: Placebo plus cognitive behavior therapy (CBT).
- Regular Sertraline Titration Plus CBT: Regular titration of sertraline (RegSert) plus cognitive behavior therapy. The titration schedule used a flexible upward titration from 25 mg/day to 200 mg/day over 9 weeks unless higher doses were not tolerated, after which the dosage was adjusted as a function of tolerability. If tolerated, maximum dose could be achieved in 5 weeks.
- Slow Sertraline Titration Plus CBT: Slow titration of sertraline (SloSert)plus cognitive behavior therapy. The titration schedule utilized a slower titration schedule relative to the RegSert arm. Unless unable to tolerate higher doses, children remained on 25mg/day for the first two weeks, 50mg/day from weeks 3-4, 75mg/day for weeks 5-6, 100mg/day for week 7, 150mg/day for week 8, and 200mg/day for week 9 until the end of the study.
Period: Overall Study
Arm/Group | Placebo Plus CBT | Regular Sertraline Titration Plus CBT | Slow Sertraline Titration Plus CBT
Started | 18 | 17 | 21
Completed | 14 | 10 | 13
Not Completed | 4 | 7 | 8
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Temporary study suspension | 2 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo plus cognitive behavior therapy.
- Regular Titration: Regular titration of sertraline plus cognitive behavior therapy.
- Slow Titration: Slow titration of sertraline plus cognitive behavior therapy.
- Total: Total of all reporting groups
Arm/Group | Placebo | Regular Titration | Slow Titration | Total
Number analyzed (Participants) | 18 | 17 | 21 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 17 | 21 | 56
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 22
  Male | 11 | 10 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Severity of Activation (CGI-SA)
Description: The CGI-SA was adapted from the Clinical Global Impressions - Severity of Illness (CGI-SI) rating (Guy, 1976). The CGI-SI is commonly used in clinical studies of children and adults and has been extensively validated (Zaider et al., 2003). On the CGI-SA clinicians rate the severity of activation symptoms on a range from 0 (no activation) to 7 (extremely severe symptoms, functionally highly impaired and/or extreme distress). We report values representing Median+/-Std Dev for the maximum CGI-SA obtained over the course of study.
Time Frame: Measured at screening, baseline and weekly until end of week 8 after baseline, then monthly for two months and finally at end of study
Population: Per protocol, Intent to treat
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Regular Titration | Slow Titration
Number analyzed (Participants) | 18 | 17 | 21
units on a scale | .50 (1.50) | 2.00 (1.35) | 2.00 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Regular Titration vs Slow Titration; Data were analyzed using two-sided Kruskal-Wallis test with level of significance = .05. Null hypothesis was that there were no group differences. The maximum CGI-SA obtained over course of study was the outcome measure; Test type: Superiority or Other; p = .2106, Kruskal-Wallis

2. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) Total Score
Description: The CY-BOCS (Scahill et al., 1997) is a semi-structured, clinician rated instrument to measure OCD symptom severity in youth. The CY-BOCS contains a symptom checklist and a severity scale. Through the symptom checklist the clinician assesses current and past experiences of over 60 potential obsessions and compulsions. The Total Score represents the sum of obsession severity and compulsion severity which each consist of five clinician ratings on a Likert scale (range from 0 (none) to 4 (extreme), for time spent, interference, distress, resistance and control over symptoms). Summing of obsession and compulsion severity (range 0-20 on each) produces the Total CY-BOCS score (range 0-40, with 0 representing the best and 40 the worst outcome). Studies have documented good psychometric properties of the CY-BOCS (Gallant et al., 2008; Scahill et al., 1997; Storch et al., 2004).
Time Frame: Measured at Week 18 or End of Study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Regular Titration: Regular titration of sertraline plus cognitive behavior therapy. The titration schedule used a flexible upward titration from 25 mg/day to 200 mg/day over 9 weeks unless higher doses were not tolerated, after which the dosage was adjusted as a function of tolerability. If tolerated, maximum dose could be achieved in 5 weeks.
Arm/Group | Placebo | Regular Titration | Slow Titration
Number analyzed (Participants) | 18 | 17 | 21
units on a scale | 16.28 (7.11) | 16.35 (9.60) | 17.67 (7.28)
Statistical Analysis 1: Comparison: Placebo vs Regular Titration vs Slow Titration; Data were analyzed using ANCOVA modeling with two-sided testing and level of significance = .05. The dependent variable was last measured CY-BOCS score, the independent variable was randomized group assignment and the covariate was the CY-BOCS score at baseline. The null hypothesis was that there were no group differences; Test type: Superiority or Other; p = .8831, ANCOVA

ADVERSE EVENTS:
Time Frame: For individual study participants Adverse Events were collected from point of informed consent to end of study (up to 19 weeks plus required wash-out periods for completers). For the entire study adverse events were collected from 2/09 to 2/11.
Arm/Group | Placebo | Regular Titration | Slow Titration
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/17 | 0/21
Other Adverse Events (participants affected / at risk) | 11/18 | 12/17 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Regular Titration (N=17) | Slow Titration (N=21)
Depersonalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Regular Titration (N=17) | Slow Titration (N=21)
Insomnia (Nervous system disorders) | 3 (10) | 8 (12) | 6 (8)
Headache (Nervous system disorders) | 9 (12) | 9 (24) | 12 (27)
diarrhea (Gastrointestinal disorders) | 2 (3) | 5 (8) | 8 (14)

LIMITATIONS AND CAVEATS:
Temporary study suspension led to smaller number of subjects enrolled than initially planned and resulted in smaller number of subjects analyzed, reducing power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No